CLINICAL TRIAL: NCT01480128
Title: A Multicenter Prospective Randomized Clinical Trail on the Efficacy of the Single Port Laparoscopic Surgery Compared With Multiport Laparoscopic Surgery
Brief Title: Multicenter Single-port Colectomy RCT
Acronym: SIMPLE
Status: Approved for marketing | Type: Expanded Access
Sponsor: The Catholic University of Korea (Other)
Collaborators: Kyunghee University (Other); Chonnam National University (Other)
Responsible Party: Principal Investigator, Hyung-Jin Kim, MD, PhD, The Catholic University of Korea
Other Study IDs: SPA-2011
Record Dates: First submitted 2011-11-23; First posted 2011-11-28 (Estimated); Last update posted 2020-06-19 (Actual); Status verified 2020-06

CONDITIONS: Colon Neoplasms
Keywords: Single-port; Laparoscopy; colectomy; Single port; colon cancer; minimally invasive surgery
MeSH Terms: conditions — Colonic Neoplasms | interventions — Laparoscopy

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Procedure: Single-port — Single-port laparoscopic colon resection
  Other Names: Single-incision; SILS; Octoport
Procedure: Multi-port — Multi-port laparoscopic colon resection
  Other Names: laparoscopy

SUMMARY:
This clinical trial is going to compare the single-port and multi-port laparoscopic colectomy for colon cancer treatment, in terms of safety, efficacy, and cost.

The investigators hypothesize that the single-port laparoscopic colectomy is not inferior to multiport laparoscopic colectomy.

DETAILED DESCRIPTION:
This clinical trial is a multicenter prospective randomized trial to compare the single-port and multi-port laparoscopic colectomy for colon cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

* colon adenocarcinoma
* curative resection
* age : 20 ~ 85

Exclusion Criteria:

* distal transverse colon cancer
* splenic flexure colon cancer
* descending colon cancer
* emergency operation
* obstruction
* perforation
* ASA 3 or 4
* pregnant woman
* tumor associated with FAP, HNPCC, or IBD
* distant metastasis
* adjacent organ invasion
* synchronous colorectal cancer
* other malignancy within last five years

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Jun-Gi Kim, MD, Principal Investigator — The Catholic University of Korea
Locations (1):
- St. Vincent's hospital, Suwon, South Korea

REFERENCES:
- [Derived] Kang BM, Lee YS, Kim JH, Kim HJ, Lee SC, Kim CW, Lim SW, Kim JG, Lee SH. Quality of life and patient satisfaction after single- and multiport laparoscopic surgery in colon cancer: a multicentre randomised controlled trial (SIMPLE Trial). Surg Endosc. 2021 Nov;35(11):6278-6290. doi: 10.1007/s00464-020-08128-9. Epub 2020 Nov 3. PMID 33141277
- [Derived] Lee YS, Kim JH, Kim HJ, Lee SC, Kang BM, Kim CW, Lim SW, Lee SH, Kim JG. Short-term Outcomes of Single-port Versus Multiport Laparoscopic Surgery for Colon Cancer: The SIMPLE Multicenter Randomized Clinical Trial. Ann Surg. 2021 Feb 1;273(2):217-223. doi: 10.1097/SLA.0000000000003882. PMID 32209897
- [Derived] Kang BM, Kim HJ, Kye BH, Lee SC, Lee KY, Park SJ, Lee SH, Lim SW, Lee YS, Kim JH, Lee J, Kim MK, Kim JG. Multicenter, randomized single-port versus multiport laparoscopic surgery (SIMPLE) trial in colon cancer: an interim analysis. Surg Endosc. 2018 Mar;32(3):1540-1549. doi: 10.1007/s00464-017-5842-0. Epub 2017 Sep 15. PMID 28916955